CLINICAL TRIAL: NCT02318303
Title: A Double-blind, Randomized, Parallel-group, Comparative Study to Evaluate the Efficacy, Safety and Tolerability of Two Different Strengths and Regimens of a Fixed Dose Combination GSP 301 Nasal Spray Compared With Placebo Nasal Spray and Individual Monotherapy Formulations (Comparators), in Subjects (12 Years of Age and Older) With Seasonal Allergic Rhinitis (SAR)
Brief Title: To Study GSP 301 in Patients With Seasonal Allergic Rhinitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Glenmark Pharmaceuticals Ltd. India (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GPL/CT/2014/004/II; IND Number: 123164 (Other: Center for Drug Evaluation and Research (CDER)); Study Number (GSP 301-201) (Other: Glenmark Pharmaceuticals Ltd.)
Record Dates: First submitted 2014-12-03; First posted 2014-12-17 (Estimated); Results first posted 2017-06-28 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-09

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — BID protein, human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (7):
- GSP 301 Placebo NS (Placebo Comparator)
  Interventions: Drug: GSP 301 Placebo NS
- GSP 301-1 NS (QD) (Experimental)
  Interventions: Drug: GSP 301-1 NS (QD)
- GSP 301-2 NS (BID) (Experimental)
  Interventions: Drug: GSP 301-2 NS (BID)
- Olopatadine HCl-1 NS (QD) (Active Comparator)
  Interventions: Drug: Olopatadine HCl-1 NS (QD)
- Olopatadine HCl-2 NS (BID) (Active Comparator)
  Interventions: Drug: Olopatadine HCl-2 NS (BID)
- Mometasone Furoate-1 NS (QD) (Active Comparator)
  Interventions: Drug: Mometasone Furoate-1 NS (QD)
- Mometasone Furoate-2 NS (BID) (Active Comparator)
  Interventions: Drug: Mometasone Furoate-2 NS (BID)

INTERVENTIONS:
Drug: GSP 301-1 NS (QD) — GSP 301-1 NS (665 μg olopatadine hydrochloride/50 μg mometasone furoate) administered as 2 sprays/nostril
  Arms: GSP 301-1 NS (QD)
Drug: GSP 301-2 NS (BID) — GSP 301-2 NS (665 μg olopatadine hydrochloride/25 μg mometasone furoate) administered as 2 sprays/nostril
  Arms: GSP 301-2 NS (BID)
Drug: GSP 301 Placebo NS — GSP 301 placebo NS administered as 2 sprays/nostril
  Arms: GSP 301 Placebo NS
Drug: Olopatadine HCl-1 NS (QD) — Olopatadine HCl-1 NS (665 μg) administered as 2 sprays/nostril
  Arms: Olopatadine HCl-1 NS (QD)
Drug: Olopatadine HCl-2 NS (BID) — Olopatadine HCl-2 NS (665 μg) administered as 2 sprays/nostril
  Arms: Olopatadine HCl-2 NS (BID)
Drug: Mometasone Furoate-1 NS (QD) — Mometasone furoate -1 NS (50 μg) administered as 2 sprays/nostril
  Arms: Mometasone Furoate-1 NS (QD)
Drug: Mometasone Furoate-2 NS (BID) — Mometasone furoate-2 NS (25 μg) administered as 2 sprays/nostril
  Arms: Mometasone Furoate-2 NS (BID)

SUMMARY:
Study to evaluate the two different strengths and dose regimen of GSP 301 to be effective in treatment of seasonal allergic rhinitis.

ELIGIBILITY:
Key Inclusion Criteria:

1. Aged ≥12 years and older inclusive of either sex.
2. Documented clinical history of SAR (for at least 2 years preceding the Screening Visit [Visit 1]) with exacerbations (clinical evidence of active symptoms) during the study season for the mountain cedar pollen
3. A 12-hour reflective TNSS ≥ 8 out of a possible 12 and a congestion score of ≥ 2 for the AM assessment at the Screening Visit (Visit 1).

Key Exclusion Criteria:

1. Pregnant or lactating women.
2. Plans to travel outside the known pollen area for the investigative site for > 24 hours during the last 7 days of run in period.
3. History of nasal polyps of other clinically significant respiratory tract malformations, recent nasal biopsy, nasal trauma (such as nasal piercing) or surgery, atopic dermatitis or rhinitis medicamentosa.
4. History of anaphylaxis and/or other severe local reaction(s) to skin testing.
5. History of positive test for HIV, Hepatitis B or Hepatitis C infection.
6. Documented evidence of acute or significant chronic sinusitis or chronic purulent postnasal drip.
7. Subjects with an active pulmonary disorder or infection.
8. Subjects with posterior subcapsular cataracts or glaucoma.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1111 (Actual)
Dates: Start 2014-12; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sudeesh Tantry, Ph.D, Study Director — Glenmark Pharmaceuticals Ltd
Locations (10):
- United States (10):
  - Glenmark Investigational Site 10, Austin, Texas
  - Glenmark Investigational Site 5, Austin, Texas
  - Glenmark Investigational Site 6, Austin, Texas
  - Glenmark Investigational Site 2, Kerrville, Texas
  - Glenmark Investigational Site 7, New Braunfels, Texas
  - Glenmark Investigational Site 3, San Antonio, Texas
  - Glenmark Investigational Site 4, San Antonio, Texas
  - Glenmark Investigational Site 8, San Antonio, Texas
  - Glenmark Investigational Site 9, San Antonio, Texas
  - Glenmark Investigational Site 1, Waco, Texas

REFERENCES:
- [Derived] Andrews CP, Mohar D, Salhi Y, Tantry SK. Efficacy and safety of twice-daily and once-daily olopatadine-mometasone combination nasal spray for seasonal allergic rhinitis. Ann Allergy Asthma Immunol. 2020 Feb;124(2):171-178.e2. doi: 10.1016/j.anai.2019.11.007. Epub 2019 Nov 15. PMID 31734334

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at 10 sites in the US.
Groups:
- Mometasone Furoate-1 NS (QD): Mometasone furoate-1 NS (50 μg) administered as 2 sprays/nostril
Period: Overall Study
Arm/Group | GSP 301 Placebo NS | GSP 301-1 NS (QD) | Mometasone Furoate-1 NS (QD) | Olopatadine HCl-1 NS (QD) | GSP 301-2 NS (BID) | Mometasone Furoate-2 NS (BID) | Olopatadine HCl-2 NS (BID)
Started | 159 | 158 | 160 | 158 | 157 | 159 | 160
Completed | 155 | 155 | 157 | 155 | 152 | 153 | 158
Not Completed | 4 | 3 | 3 | 3 | 5 | 6 | 2

BASELINE CHARACTERISTICS:
Groups:
- GSP 301-1 NS (QD): GSP 301-1 NS administered as 2 sprays/nostril
- Mometasone Furoate-1 NS (QD): Mometasone furoate-1 NS administered as 2 sprays/nostril
- Olopatadine HCl-1 NS (QD): Olopatadine HCl-1 NS administered as 2 sprays/nostril
- GSP 301-2 NS (BID): GSP 301-2 NS administered as 2 sprays/nostril
- Mometasone Furoate-2 NS (BID): Mometasone furoate-2 NS administered as 2 sprays/nostril
- Olopatadine HCl-2 NS (BID): Olopatadine HCl-2 NS administered as 2 sprays/nostril
- Total: Total of all reporting groups
Arm/Group | GSP 301 Placebo NS | GSP 301-1 NS (QD) | Mometasone Furoate-1 NS (QD) | Olopatadine HCl-1 NS (QD) | GSP 301-2 NS (BID) | Mometasone Furoate-2 NS (BID) | Olopatadine HCl-2 NS (BID) | Total
Number analyzed (Participants) | 159 | 158 | 160 | 158 | 157 | 159 | 160 | 1111
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.35 (14.951) | 43.83 (13.609) | 44.40 (14.312) | 41.90 (12.478) | 43.44 (14.128) | 44.58 (13.698) | 43.49 (13.868) | 43.86 (13.882)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 112 | 100 | 115 | 105 | 111 | 96 | 101 | 740
  Male | 47 | 58 | 45 | 53 | 46 | 63 | 59 | 371

OUTCOME MEASURES:

1. Primary Outcome: Change in rTNSS From Baseline to End of Treatment
Description: Subjects were asked to assess rTNSS (reflective Total Nasal Symptom Score), ie, an evaluation of symptom severity over the past 12 hours prior to the recording of the score. The TNSS was defined as the sum of the subject-reported symptom severity scores for the following four nasal symptoms, recorded by each subject in the diary: rhinorrhea, sneezing, nasal congestion, nasal itching.
  The total rTNSS scores for all four symptoms (i.e, the lowest possible score (0) and the highest possible score (12).) Higher score means a worse outcome.
  The severity scale for each symptom evaluation was defined as follows:
  * 0 = absent (no sign/symptom evident)
  * 1 = mild (sign/symptom clearly present, but minimal awareness; easily tolerated)
  * 2 = moderate (definite awareness of sign/symptom that is bothersome but tolerable)
  * 3 = severe (sign/symptom that is hard to tolerate [i.e., causes interference with activities of daily living and/or sleeping])
Time Frame: 14 days
Population: The full analysis set (FAS) included all randomized subjects who received at least one dose of randomized study medication and had at least one post-baseline primary efficacy assessment. This was the primary analysis set for efficacy analyses.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- GSP 301 Placebo: GSP 301 placebo NS administered as 2 sprays/nostril
- GSP 301-1 NS (QD): GSP 301-1 NS (QD) administered as 2 sprays/nostril
- Mometasone Furoate-1 NS (QD): Mometasone furoate-1 NS (QD) administered as 2 sprays/nostril
- Olopatadine HCl-1 NS (QD): Olopatadine HCl-1 NS (QD) administered as 2 sprays/nostril
- GSP 301-2 NS (BID): GSP 301-2 NS (BID) administered as 2 sprays/nostril
- Mometasone Furoate-2 NS (BID): Mometasone furoate-2 NS (BID) administered as 2 sprays/nostril
- Olopatadine HCl-2 NS (BID): Olopatadine HCl-2 NS (BID) administered as 2 sprays/nostril
Arm/Group | GSP 301 Placebo | GSP 301-1 NS (QD) | Mometasone Furoate-1 NS (QD) | Olopatadine HCl-1 NS (QD) | GSP 301-2 NS (BID) | Mometasone Furoate-2 NS (BID) | Olopatadine HCl-2 NS (BID)
Number analyzed (Participants) | 158 | 158 | 160 | 158 | 157 | 159 | 160
units on a scale
  Baseline | 10.3 (1.18) | 10.4 (1.24) | 10.4 (1.30) | 10.3 (1.26) | 10.4 (1.19) | 10.5 (1.13) | 10.3 (1.24)
  Change from Baseline to Visit 4 | -1.4 (2.00) | -2.5 (2.52) | -2.2 (2.68) | -1.7 (2.09) | -2.6 (2.56) | -1.9 (1.88) | -2.1 (2.26)
Statistical Analysis 1: Comparison: GSP 301 Placebo vs GSP 301-1 NS (QD); Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -1.1087, 97.5% CI 2-sided [-1.6690 to -0.5485]
Statistical Analysis 2: Comparison: GSP 301 Placebo vs GSP 301-2 NS (BID); Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -1.1703, 97.5% CI 2-sided [-1.7315 to -0.6090]
Statistical Analysis 3: Comparison: GSP 301-1 NS (QD) vs Olopatadine HCl-1 NS (QD); Test type: Superiority; p = 0.0020, ANCOVA; Mean Difference (Final Values) = -0.7718, 95% CI 2-sided [-1.2616 to -0.2820]
Statistical Analysis 4: Comparison: GSP 301-1 NS (QD) vs Mometasone Furoate-1 NS (QD); Test type: Superiority; p = 0.1524, ANCOVA; Mean Difference (Final Values) = -0.3563, 95% CI 2-sided [-0.8445 to 0.1319]
Statistical Analysis 5: Comparison: GSP 301-2 NS (BID) vs Olopatadine HCl-2 NS (BID); Test type: Superiority; p = 0.0488, ANCOVA; Mean Difference (Final Values) = -0.4918, 95% CI 2-sided [-0.9810 to -0.0025]
Statistical Analysis 6: Comparison: GSP 301-2 NS (BID) vs Mometasone Furoate-2 NS (BID); Test type: Superiority; p = 0.0043, ANCOVA; Mean Difference (Final Values) = -0.7133, 95% CI 2-sided [-1.2031 to -0.2235]

ADVERSE EVENTS:
Time Frame: AEs and SAEs were collected from the time of signing the informed consent form until the follow-up contact
Arm/Group | GSP 301 Placebo NS | GSP 301-1 NS (QD) | Mometasone Furoate-1 NS (QD) | Olopatadine HCl-1 NS (QD) | GSP 301-2 NS (BID) | Mometasone Furoate-2 NS (BID) | Olopatadine HCl-2 NS (BID)
Serious Adverse Events (participants affected / at risk) | 0/159 | 1/158 | 0/160 | 0/158 | 0/157 | 0/159 | 0/160
Other Adverse Events (participants affected / at risk) | 0/159 | 0/158 | 0/160 | 0/158 | 0/157 | 0/159 | 0/160
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSP 301 Placebo NS (N=159) | GSP 301-1 NS (QD) (N=158) | Mometasone Furoate-1 NS (QD) (N=160) | Olopatadine HCl-1 NS (QD) (N=158) | GSP 301-2 NS (BID) (N=157) | Mometasone Furoate-2 NS (BID) (N=159) | Olopatadine HCl-2 NS (BID) (N=160)
Gastrointestinal ulcer and Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — There were two SAEs (gastrointestinal ulcer and gastritis) reported both in the same subject.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Per the agreement, Sponsor reserves the right for publishing trial results and the Investigator cannot publish without written consent from the CRO/ Sponsor.